CLINICAL TRIAL: NCT01334749
Title: Determinants of Dementia After Stroke
Brief Title: Observational Study on Determinants of Dementia After Stroke
Acronym: DEDEMAS
Status: Active, not recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Martin Dichgans, Prof. Dr. med. M. Dichgans, Ludwig-Maximilians - University of Munich
Other Study IDs: ISD-DEDEMAS-01
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: Stroke; Dementia; Dementia, Vascular; Alzheimer's Disease; Intracranial Hemorrhage; Brain Ischemia
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke; Dementia; Dementia, Vascular; Alzheimer Disease; Intracranial Hemorrhages; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, RNA, CSF
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Stroke: Patients over 18 years and without pre-stroke dementia, displaying an ischemic or hemorrhagic stroke, onset within the last 72 hours, language German

SUMMARY:
The primary aim of the DEDEMAS (Determinants of Dementia After Stroke) study is to identify predictors of post stroke dementia (PSD). A particular focus will be on biological markers (neuroimaging, biochemical markers derived from blood) and on interactions between vascular and neurodegenerative mechanisms. For this purpose patients with an acute stroke and without prior dementia will be followed for 10 years.

Note: Starting from 01.01.2014 this study is expanded to a multi-centric design funded by the German Center for Neurodegenerative Diseases (The DZNE - Mechanisms of Dementia After Stroke (DEMDAS) Study). This includes the following study sites: DZNE/München - Institute for Stroke and Dementia Research, Klinikum der Universität München (Coordinator); DZNE/Berlin - Neuroscience Research Center - Campus Mitte Charité; DZNE/Bonn - Klinik und Poliklinik für Neurologie, Universitätsklinikum Bonn; DZNE/Göttingen - University Medical Center Göttingen; DZNE/Magdeburg - Universitätsklinikum Magdeburg.

DETAILED DESCRIPTION:
Risk of dementia is high after stroke but the mechanisms of post stroke dementia (PSD) are insufficiently understood. Specifically, there are few data on how vascular and neurodegenerative mechanisms interact in determining cognitive decline after stroke. The primary aim of the DEDEMAS/DEMDAS (Determinants of Dementia After Stroke) study is to identify predictors of PSD. A particular focus will be on biological markers (neuroimaging, biochemical markers derived from blood) and on interactions between vascular and neurodegenerative mechanisms. Patients with an acute stroke and without prior dementia will be followed for 5 years with assessments at baseline (< 72 h after onset of stroke), and at 3, 6, 12, 24, 36, 48, and 60 months. In addition, DEDEMAS patients will have an annual telephone follow-up from year 6 to 10. Baseline assessments will include variables previously demonstrated to be associated with PSD as well as novel variables. Brain MRI (structural MRI and resting state fMRI) in combination with detailed neuropsychological testing and blood draws will be done at 6, 12, 36, and 60 months. Patients developing cognitive impairment (with or without dementia) and a subgroup of matched individuals without cognitive decline will be examined by brain FDG-PET and Amyloid-PET scanning. Lumbar puncture will be done on patients who develop cognitive impairment and thus have a clinical indication for the procedure. Efforts will be made to classify demented patients into diagnostic categories (Vascular Dementia, Mixed Dementia, Alzheimer's disease, other categories). Predictive factors for PSD will be identified using multiple Cox-proportional hazards models. Apart from providing insights into the mechanisms of PSD this study holds the potential to identify novel diagnostic markers and novel targets for preventive therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Language: German
* Acute stroke that occurred within the last 5 days as defined by:

acute focal neurological deficit in combination with one of the following:

* An acute ischemic infarct as documented by either a DWI positive lesion on MR imaging or a new lesion on a delayed CT scan
* An intracerebral hemorrhage as documented on CT or MRI
* An informant of the patient is available
* Written informed consent by patient prior to study participation
* Willingness to participate in follow-up

Exclusion Criteria:

* IQCODE > 64 or diagnosis of dementia
* Patients transferred from an outside stroke unit (to avoid possible selection bias)
* Patients presenting a stroke going back more than 120 hours
* Patients presenting one of the following diseases: cerebral venous thrombosis, traumatic cerebral haemorrhage, intracerebral haemorrhage because of a known or image-guided assumed vascular malformation, pure meningeal or intraventricular haemorrhage
* Patients presenting a malignant disease with life expectancy < 3years
* Contraindication for MRI
* Participation in an intervention/AMG-study at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a specialized stroke service because of an acute stroke.
Sampling Method: Probability Sample
Enrollment: 736 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
dementia occurrence | 5 years in DEMDAS
  this evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the instrumental activities daily life scale after an interview with the patient and his/her family
dementia occurrence | 10 years in DEDEMAS
  this evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the instrumental activities daily life scale after an interview with the patient and his/her family

SECONDARY OUTCOMES:
dementia occurrence | 6 months
  this evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the instrumental activities daily life scale after an interview with the patient and his/her family
dementia occurrence | 12 months
  this evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the instrumental activities daily life scale after an interview with the patient and his/her family
dementia occurrence | 36 months
  this evaluation will be based on a neurological and general clinical examination, and on the evaluation of activities of daily life using the instrumental activities daily life scale after an interview with the patient and his/her family
cognitive impairment | 6 months
  Impairment of some tests of cognitive battery without significant impairment in activities of daily living
cognitive impairment | 12 months
  Impairment of some tests of cognitive battery without significant impairment in activities of daily living
cognitive impairment | 36 months
  Impairment of some tests of cognitive battery without significant impairment in activities of daily living
cognitive impairment | 60 months
  Impairment of some tests of cognitive battery without significant impairment in activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dichgans, Prof., Principal Investigator — Institute for Stroke and Dementia Research, Klinikum der Universität München
Locations (5):
- Germany (5):
  - DZNE/Munich-Interdisciplinary Stroke Center Munich, Klinikum der Universität München, Campus Großhadern, Munich, Bavaria
  - DZNE/Berlin - Neuroscience Research Center - Campus Mitte Charité, Berlin
  - DZNE/Bonn - Klinik und Poliklinik für Neurologie, Universitätsklinikum Bonn, Bonn
  - DZNE/Göttingen - University Medical Center Göttingen, Göttingen
  - DZNE/Magdeburg - Universitätsklinikum Magdeburg, Magdeburg

REFERENCES:
- [Background] Wollenweber FA, Zietemann V, Rominger A, Opherk C, Bayer-Karpinska A, Gschwendtner A, Coloma Andrews L, Burger K, Duering M, Dichgans M. The Determinants of Dementia After Stroke (DEDEMAS) Study: protocol and pilot data. Int J Stroke. 2014 Apr;9(3):387-92. doi: 10.1111/ijs.12092. Epub 2013 Jul 9. PMID 23834337
- [Result] Wollenweber FA, Darr S, Muller C, Duering M, Buerger K, Zietemann V, Malik R, Brendel M, Ertl-Wagner B, Bartenstein P, Rominger A, Dichgans M. Prevalence of Amyloid Positron Emission Tomographic Positivity in Poststroke Mild Cognitive Impairment. Stroke. 2016 Oct;47(10):2645-8. doi: 10.1161/STROKEAHA.116.013778. Epub 2016 Aug 18. PMID 27539301
- [Result] Zietemann V, Kopczak A, Muller C, Wollenweber FA, Dichgans M. Validation of the Telephone Interview of Cognitive Status and Telephone Montreal Cognitive Assessment Against Detailed Cognitive Testing and Clinical Diagnosis of Mild Cognitive Impairment After Stroke. Stroke. 2017 Nov;48(11):2952-2957. doi: 10.1161/STROKEAHA.117.017519. Epub 2017 Oct 17. PMID 29042492
- [Result] von Rennenberg R, Nolte CH, Liman TG, Hellwig S, Riegler C, Scheitz JF, Georgakis MK, Fang R, Bode FJ, Petzold GC, Hermann P, Zerr I, Goertler M, Bernkopf K, Wunderlich S, Dichgans M, Endres M; DEMDAS investigators *. High-Sensitivity Cardiac Troponin T and Cognitive Function Over 12 Months After Stroke-Results of the DEMDAS Study. J Am Heart Assoc. 2024 Mar 19;13(6):e033439. doi: 10.1161/JAHA.123.033439. Epub 2024 Mar 8. PMID 38456438
- [Result] Georgakis MK, Fang R, During M, Wollenweber FA, Bode FJ, Stosser S, Kindlein C, Hermann P, Liman TG, Nolte CH, Kerti L, Ikenberg B, Bernkopf K, Poppert H, Glanz W, Perosa V, Janowitz D, Wagner M, Neumann K, Speck O, Dobisch L, Duzel E, Gesierich B, Dewenter A, Spottke A, Waegemann K, Gortler M, Wunderlich S, Endres M, Zerr I, Petzold G, Dichgans M; DEMDAS Investigators. Cerebral small vessel disease burden and cognitive and functional outcomes after stroke: A multicenter prospective cohort study. Alzheimers Dement. 2023 Apr;19(4):1152-1163. doi: 10.1002/alz.12744. Epub 2022 Jul 25. PMID 35876563
- [Derived] Arlt FA, Sperber PS, von Rennenberg R, Gebert P, Teegen B, Georgakis MK, Fang R, Dewenter A, Gortler M, Petzold GC, Wunderlich S, Zerr I, Dichgans M, Pruss H, Endres M; DEMDAS Investigators. Serum anti-NMDA receptor antibodies are linked to memory impairment 12 months after stroke. Mol Psychiatry. 2025 Apr;30(4):1359-1368. doi: 10.1038/s41380-024-02744-w. Epub 2024 Oct 30. PMID 39478168
- [Derived] Duering M, Adam R, Wollenweber FA, Bayer-Karpinska A, Baykara E, Cubillos-Pinilla LY, Gesierich B, Araque Caballero MA, Stoecklein S, Ewers M, Pasternak O, Dichgans M. Within-lesion heterogeneity of subcortical DWI lesion evolution, and stroke outcome: A voxel-based analysis. J Cereb Blood Flow Metab. 2020 Jul;40(7):1482-1491. doi: 10.1177/0271678X19865916. Epub 2019 Jul 25. PMID 31342832
- See also: Related Info — http://www.klinikum.uni-muenchen.de/Interdisziplinaeres-Schlaganfallzentrum/en/index.html
- See also: Related Info — http://www.klinikum.uni-muenchen.de/Institut-fuer-Schlaganfall-und-Demenzforschung/en/index.html